CLINICAL TRIAL: NCT02734420
Title: Effect of Photodynamic Therapy With Low-level Laser on Infected Dentin in Primary Teeth: A Controlled Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Zenildo Santos Silva Jr., D.D.S, M.Sc.Ph.D, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZENILDOJUNIOR
Record Dates: First submitted 2013-09-13; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Dental Caries
Keywords: Dental caries; PDT; LLLT; pediatric dentistry
MeSH Terms: conditions — Dental Caries | interventions — 1-phenyl-3,3-dimethyltriazene; Photochemotherapy; Tolonium Chloride; Lasers

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PapacarieMBlue and PDT (Experimental): Initial periapical and interproximal radiographs; Microbiological sample with otoscope curette to standardize volume of carious tissue; Application on PapacarieMBlue (addition of toluidine blue) for 5 minutes to potentiate effect of PDT; Removal of carious tissue around lateral walls of the cavity with non-cutting curette; No removal of carious tissue on pulp floor; Irradiation of dental tissue for one minute on a single point; Second microbiological sample of remaining dentin with curette; Restoration with glass ionomer cement (Ketac Molar EasyMIx 3M ESPE); Follow up: Radiographic control: periapical and interproximal radiographs at 3, 6 and 12 months.
  Interventions: Drug: PapacarieMBlue and PDT; Device: Laser
- Toluidine Blue O and PDT (Experimental): Initial periapical and interproximal radiographs;Microbiological sample with otoscope curette to standardize volume of carious tissue;Application of Toluidine Blue O for 5 minutes to potentiate effect of PDT; Removal of carious tissue around lateral walls of the cavity with sharp curette; No removal of carious tissue on pulp floor;non-cutting curette; Irradiation of dental tissue for one minute on a single point;Second microbiological sample of remaining dentin with curette; Follow up; Radiographic control: periapical and interproximal radiographs at 3, 6 and 12 months.
  Interventions: Drug: Toluidine Blue O and PDT; Device: Laser

INTERVENTIONS:
Drug: PapacarieMBlue and PDT — Initial periapical and interproximal radiographs Microbiological sample with otoscope curette to standardize volume of carious tissue; Application on PapacarieMBlue (addition of toluidine blue) for 5 minutes to potentiate effect of PDT; Removal of carious tissue around lateral walls of the cavity with non-cutting curette; No removal of carious tissue on pulp floor; Irradiation of dental tissue for one minute on a single point; Second microbiological sample of remaining dentin with curette; Clinical evaluation by inspection of texture of remaining dentin with exploratory probe; Restoration with glass ionomer cement (Ketac Molar EasyMIx 3M ESPE); Follow up;Radiographic control: periapical and interproximal radiographs at 3, 6 and 12 months.
  Other Names: Photodynamic therapy and lower level laser therapy
  Arms: PapacarieMBlue and PDT
Drug: Toluidine Blue O and PDT — Initial periapical and interproximal radiographs;Microbiological sample with otoscope curette to standardize volume of carious tissue;Application of Toluidine Blue O for 5 minutes to potentiate effect of PDT; Removal of carious tissue around lateral walls of the cavity with sharp curette; No removal of carious tissue on pulp floor;non-cutting curette; Irradiation of dental tissue for one minute on a single point;Second microbiological sample of remaining dentin with curette;Clinical evaluation by inspection of texture of remaining dentin with exploratory probe; Restoration with glass ionomer cement (Ketac Molar EasyMIx 3M ESPE);Follow up;Radiographic control: periapical and interproximal radiographs at 3, 6 and 12 months.
  Other Names: Photodynamic therapy and lower level laser therapy
  Arms: Toluidine Blue O and PDT
Device: Laser

SUMMARY:
The aim of the proposed study is to assess the clinical effect of photodynamic therapy (PDT) on dentin with carious lesions in primary teeth. Patients with primary molars exhibiting deep carious lesions on the occlusal surface indicated for restorative treatment will be randomly allocated to three groups: Group 1 - traditional caries removal with a low-speed drill; Group 2 - PDT + PapaMblue (carious tissue removal agent) modified with methylene blue; and Group 3 - PDT with methylene blue 0.05%. PDT will be performed with low-level laser for the treatment of the carious tissue. Dentin samples will be removed before and after PDT for microbiological analysis. The microbiological samples will be cultured in Brucella blood agar, Mitis Salibarius-bacitracin agar and Rogosa SL agar. The teeth will then be restored using high-viscosity glass ionomer cement, with clinical and radiographic follow up at six, 12 and 24 months. The data will be submitted to descriptive statistics.

DETAILED DESCRIPTION:
The groups of study (Group 1)- Conventional caries removal with low-speed drill (Group 2)- PDT combined with PapaMblue (Group 3)- PDT combined with methylene blue

The data in descriptive statistics will be used The chi-squared test and Fisher's exact test will be used for the comparison of categorical variables (age and gender). The Student's t-test and analysis of variance will be used for the comparison of signs and symptoms of reversible pulpitis. Pearson's correlation coefficients will be calculated to determine the strength of correlations among the continuous variables.

ELIGIBILITY:
Inclusion Criteria:

Adequate health, with no systemic conditions; Cooperative behavior; Presence of at least one primary molar with acute, active carious lesion not surpassing 2/3 of the dentin and only involving the occlusal face, with direct view and access and no clinical or radiographic signs of pulp involvement

Exclusion Criteria:

Systemic condition; Uncooperative behavior; Class II, III, IV or V carious lesion (Black's classification); Clinical evidence of carious lesion involving enamel, deficient restorations, insufficient size of carious lesion on dentin for access to dental instrument, hidden carious lesions, sign or symptom of pulp involvement, clinical impossibility of restoration; Radiographic evidence of pulp involvement; carious lesion surpassing 2/3 of dentin.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Microbiological analysis - collection of dentinal tissue and restoration with glass ionomer cement | 24 months
  Based on a study by Guglielmi et al. (2011)(30) teeth with be selected (n = 48) and divided into three groups, as delineated in Chart 4. Fragments of dentinal tissue will be collected from all teeth before and after treatment for microbiological analysis. The teeth will be restored with glass ionomer cement in all cases.

SECONDARY OUTCOMES:
Radiographs evaluation | up to 24 mounth
  Radiographic subtraction and the evaluation of the density of the remaining dentin will be performed prior to and following treatment for the removal of carious tissue as well as at six, 12 and 24 months after treatment. Periapical radiographs will be performed initially to include or exclude teeth based on the eligibility criteria. Immediately following the clinical procedure, the first bitewing radiograph will be taken. Bitewing x-rays will also be taken during the three follow up sessions.The bitewing x-rays will be standardized using a positioner. A portion of self-curing acrylic resin will be placed on the surface of the tooth to be evaluated and its antagonist for the impression of the surface anatomy and adapted to the positioner. This will allow the same positioning of the film during the different evaluations as well as the standardization of the x-rays at the same vertical and horizontal angles and distance for all radiographs taken with the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Bussadori, Dentist, Study Director — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costa-Santos L, Silva-Junior ZS, Sfalcin RA, Mota ACCD, Horliana ACRT, Motta LJ, Mesquita-Ferrari RA, Fernandes KPS, Prates RA, Silva DFT, Deana A, Bussadori SK. The effect of antimicrobial photodynamic therapy on infected dentin in primary teeth: A randomized controlled clinical trial protocol. Medicine (Baltimore). 2019 Apr;98(15):e15110. doi: 10.1097/MD.0000000000015110. PMID 30985667
- See also: Estudo clínico controlado do efeito da terapia fotodinâmica com laser de baixa potência em dentina infectada de dentes decíduos. — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisa.jsf